CLINICAL TRIAL: NCT03197207
Title: Quantitative Analysis of Different Acupuncture Needle Manipulation to Treat Chronic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105-0313C
Record Dates: First submitted 2017-05-11; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Lifting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lifting and thrusting (Experimental): "Dragon and Tiger warring" in lifting and thrusting
  Interventions: Procedure: "Dragon and Tiger warring" in lifting and thrusting
- twisting and rotating (Experimental): "Dragon and Tiger warring" in twisting-rotating
  Interventions: Procedure: "Dragon and Tiger warring" in twisting-rotating

INTERVENTIONS:
Procedure: "Dragon and Tiger warring" in lifting and thrusting — "Tight press" slow insert in each acupoint through the superficial,intermediate, deep layer, then "tight lifting" slow withdraw needle through the deep, intermediate, superficial layer . Two acupoints (GB34, GB39) are manipulation in the process three times each during one minute, then let patients lift shoulder up and down for three times, then draw out the needle 20 minutes later.
  Arms: lifting and thrusting
Procedure: "Dragon and Tiger warring" in twisting-rotating — When needle insert in each acupoint through the superficial,intermediate, deep layer, within each layer twisting thumb forward nine times, then twisting backward six times. Two acupoints (GB34, GB39) are manipulation in the process during one minute, then let patients lift shoulder up and down for three times, then draw out the needle 20 minutes later.
  Arms: twisting and rotating

SUMMARY:
The plan " Quantitative analysis of different acupuncture needle manipulation to treat chronic shoulder pain "includes an objective observation of acupuncture operation (movement in the form of acupuncture needles, intensity, etc.) and the body (acupoints) reactions. Patients during 20-55 years old suffered shoulder pain more than six weeks with numerical rating scale (NRS) pain intensity more than 5 points, and the previous month were not taking medicine or Western medicine were included. Then use of distal acupoints GB34 and GB39, giving once acupuncture manipulation therapy.

DETAILED DESCRIPTION:
Numerical rating scale (NRS) and pain pressure algometer were used to objective and quantitative assessment of the patient's pain. And shoulder pain and disability index-SPADI was used to objectively assess the functional changes of acupuncture treatment in patients with chronic shoulder pain. Massachusetts General Hospital Acupuncture Sensation Scale - MASS was used to get objectively record of de-qi when needle manipulation for the the body (acupoints) reactions. Acusensor2 was used to get objective observation reaction during needling manipulation, the sensor provided measurement parameters such as the lift and thrust, twisting, strength and torque during needle manipulation. Investigators will study and analysis associated clinical outcome with needling process, the needle manipulation by lifting-thrusting or twisting-rotating during the process of reinforce method or reducing method to study its dynamics and kinematics.

ELIGIBILITY:
Inclusion Criteria:

* (A) have agreed to participate in the trial and signed by the Chang Geng Memorial Hospital Human Body Test Committee approved the human test consent.
* (B) suffering from chronic shoulder pain (including frozen shoulder, or rotator cuff injury, or subclavian bursitis, Or biceps tendonitis or nonspecific shoulder pain).
* (C) at least six weeks before the screening period of shoulder pain, digital grading scale measurement of pain intensity of 5 points or more.

Exclusion Criteria:

* (A) shoulder fracture
* (B) intra-articular infection
* (C) stroke hemiplegia
* (D) spinal cord injury
* (E) postoperative shoulder surgery
* (F) pregnant woman,
* (G) took traditional Chinese medicine or Western medicine, less than one month before the screening period

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Numerical rating scale (NRS) during needle manipulation | Through study completion, an average of 5 minutes.
  Pain scale, smaller score, less pain. NRS in T0(before needle manipulation), T1(after GB34 "de-qi" ), T2(after GB34 "Dragon and Tiger warring" ), T3(after GB39 "de-qi" ), T4(after GB39 "Dragon and Tiger warring" ), T5(after Retaining Needle 20 minutes), T6(Telephone access, 24 hours later)

SECONDARY OUTCOMES:
Change in Pain pressure algometer (PA) during needle manipulation | Through study completion, an average of 5 minutes.
  The higher the score, the greater the strength that can be tolerated. PA in T0(before needle manipulation), T1(after GB34 "de-qi" ), T2(after GB34 "Dragon and Tiger warring" ), T3(after GB39 "de-qi" ), T4(after GB39 "Dragon and Tiger warring" ), T5(after Retaining Needle 20 minutes)
Change in Massachusetts General Hospital Acupuncture Sensation Scale (MASS) during needle manipulation | Through study completion, an average of 5 minutes.
  objectively measure sensation associated with 'de qi' sensation. MASS in T1(after GB34 "de-qi" ), T2(after GB34 "Dragon and Tiger warring" ), T3(after GB39 "de-qi" ), T4(after GB39 "Dragon and Tiger warring" )
Change in Shoulder Pain & Disability Index (SPADI) | Through study completion, an average of 10 minutes.
  13 items that assess two domains, 5-item subscale that measures pain, 8-item subscale that measures disability. T0(before needle manipulation), T5(after Retaining Needle 20 minutes), T6(Telephone access, 24 hours later)

OTHER OUTCOMES:
Change in Acusensor2, Needle manipulation parameters | Through study completion, an average of 5 minutes.
  Measurement of lift and thrust, twisting, strength and torque during needle manipulation. The real-time motion and force tracings records created during needle manipulation will be combined to report needling motion and force profiles pictures. Displacement (mm), Rotation (rev), Force (mN), Torque (microNm). Ta(during GB34 "Dragon and Tiger warring" ), Tb(during GB39 "Dragon and Tiger warring" )

CONTACTS AND LOCATIONS:
Overall Officials: Horng-Sheng Shiue, Dr., Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xue HS, Zhang J. [Manipulation and comprehensive application of reinforcing-reducing methods according to numbers and directions of rotation]. Zhongguo Zhen Jiu. 2013 Sep;33(9):809-13. Chinese. PMID 24298773